CLINICAL TRIAL: NCT02767973
Title: To Identify Persons Who Are Susceptible to WSP-induced Inflammation and Examine the Role of GSTM1 and Other Factors in This Susceptibility
Acronym: SmokeScreen
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: We no longer have access to the Wood smoke chamber and will need to rework how we do the wood smoke exposures.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 15-1775; 1R01ES025124-01A1 (NIH)
Record Dates: First submitted 2016-05-03; First posted 2016-05-11 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Airway Inflammation; Allergic Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Woodsmoke Exposure (Experimental)
  Interventions: Other: Wood Smoke Particles (WSP)

INTERVENTIONS:
Other: Wood Smoke Particles (WSP) — After baseline (pre-exposure) assessment (which includes recovery of induced sputum), these volunteers will then undergo an exposure to 500μg/m3 wood smoke particles for 2 hours, with alternating 15 min of exercise (cycle ergometer) with 15 min rest to achieve 25 l/m2 body surface/min minute ventilation, followed by sputum induction after 6 and 24 hours after initiation of the challenge.

SUMMARY:
Purpose: This screening protocol is designed to assess PMN (neutrophil) responsiveness to wood smoke particles (WSP) and the effect of the GSTM1 null genotype on this response. The researches will identify persons responsive and resistant to the inflammatory effect of WSP. It is anticipated that the GSTM1 genotype will be a risk factor for increased response to WSP.

DETAILED DESCRIPTION:
Particulate matter (PM) is a leading cause of respiratory tract and cardiovascular disease in the United States and world-wide. Wood smoke particles (WSP) derived from wild land and other fires account for a significant fraction of ambient air PM. Health effects associated with WSP include acute bronchitis, asthma exacerbation, pneumonia, cough and systemic inflammation. While these effects are seen in both healthy and asthmatic individuals, many studies indicate that asthmatics have increased susceptibility to the effects of WSP. Though WSP-related effects on cardiovascular (CV) disease are less well documented, WSP do contribute to PM levels, and PM exposure is linked to CV health effects (changes in heart rate variability, vascular reactivity, and lipid profiles). WSP from wild land fires can cause abrupt increases in ambient air PM 2.5 levels (mean levels ~250µg/m3, peak levels >1000 µg/m3). Avoidance of rapidly increasing PM air pollution due to wild land fires is not feasible, as many people cannot leave the burn region.

This is a screening protocol to ensure that there ultimately will be adequate subjects available for testing gamma tocopherol in an appropriate population. It will identify volunteers who have a ≥10% increase in %PMNs following WSP challenge over baseline values (SA1). This screening procedure will identify various risk factors that may increase risk of experiencing airway inflammation and related adverse health outcomes following WSP exposure. The GSTM1- genotype is a risk factor that has been extensively explored. Researchers at the CEMALB have reported that GSTM1- healthy volunteers (HVs) have increased inflammatory and systemic responses to O3 and various components of PM (LPS70 and Diesel exhaust particles). Using the 10% increase in %PMNs to define PMN responsiveness, results showed that GSTM1- volunteers had a 13 fold higher risk of being PMN responders to 0.06 ppm O3. When examining %PMNs as a continuous measure, it was observed that GSTM1- volunteers have increased airway PMN response O3 as well as increased airway and systemic PMN response to LPS70.

The researchers at the CEMALB have also examined various response features of 27 individuals (13 healthy, 4 allergic non asthmatics, 10 allergic asthmatics) defined as being responsive (R, n=18) or non-responsive (NR, n=9) to O3 based on airway PMN influx (%PMNs). Among the factors explored were inflammatory responses, baseline characteristics and gene expression profiles in recovered sputum cells. The researchers have also observed that within individuals, PMN response to O3 and LPS correlate, and anticipate that WSP will induce inflammatory responses via mechanisms similar to those for these pollutants.

ELIGIBILITY:
Inclusion Criteria

1. Age 18-45 of both genders
2. Negative pregnancy test for females who are not s/p hysterectomy with oopherectomy
3. Calculated 10 year risk of CVD by the Framingham risk score of <5%
4. Proof of Covid vaccination

Specific for Healthy Volunteers

4. No history of episodic wheezing, chest tightness or shortness of breath consistent with asthma, or physician diagnoses asthma.

5. FEV1 of at least 80% of predicted and FEV1/FVC ratio of at least .70

Specific for Allergic Asthmatic Volunteers

6. History of episodic wheezing, chest tightness, or shortness of breath consistent with asthma, or physician diagnosed asthma.

7. A POST-bronchodilator increase in FEV1 of at least 12%, OR a clinical history of asthma after the age of 6.

8. FEV1 of at least 75% of predicted without use of short acting bronchodilating medications for 12 hours, consistent with lung function of persons with no more than mild episodic or mild persistent asthma.

9. Mild persistent asthmatics must be well controlled (in accordance with NHLBI guidelines) and willing to discontinue Singulair, inhaled corticosteroids or cromolyn for a period of 2 weeks prior to study visits (except for use of cromolyn exclusively prior to exercise)

10. Allergic sensitization to at least one of the following allergen preparations: (House Dust Mite f, House dust mite p, Cockroach, Tree mix, Grass Mix, Weed Mix, Mold Mix 1, Mold Mix 2, Rat, Mouse, Guinea Pig, Rabbit, Cat or Dog) confirmed by positive immediate skin test response; or a clinical history consistent with seasonal or perennial allergy symptoms.

11. Subjects must be willing to avoid caffeine for 12 hours prior to all visits.

Allergy skin testing are performed as part of IRB98-0799, which a subject must complete in order to be considered for this protocol.

Exclusion Criteria

Patients who meet any of these criteria are not eligible for enrollment as study participants:

1. Clinical contraindications:

   1. Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, history of chronic infections/immunodeficiency, history of tuberculosis.
   2. Viral upper respiratory tract infection within 4 weeks of challenge.
   3. Any acute infection requiring antibiotics within 4 weeks of exposure or fever of unknown origin within 4 weeks of challenge.
   4. Abnormal physical findings at the baseline visit, including but not limited to abnormalities on auscultation, temperature of 37.8° C, Systolic BP > 150mm Hg or < 85 mm Hg; or Diastolic BP > 90 mm Hg or < 50 mm Hg, or pulse oximetry saturation reading less than 94%.
   5. Unwillingness to use reliable contraception if sexually active (IUD, birth control pills/patch, condoms).
   6. Use of immunosuppressive or anticoagulant medications including routine use of NSAIDS. Oral contraceptives are acceptable, as are Antidepressants and other medications may be permitted if, in the opinion of the investigator, the medication will not interfere with the study procedures or compromise safety and if the dosage has been stable for 1 month
   7. Orthopedic in juries or impediments that would preclude bicycle or treadmill exercise.
   8. Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
   9. Medications which may impact the results of the WSP exposure, interfere with any other medications potentially used in the study (to include steroids, beta antagonists, non-steroidal anti-inflammatory agents).
   10. Inability to avoid NSAIDS, Multivitamins, Vitamin C or E or herbal medications in the 4 days prior to the screening visit the exposure session.
   11. Symptomatic allergic rhinitis or current active allergies.
   12. Cigarette smoking > 1 pack per month
   13. Current symptoms of Covid infection
   14. Positive Covid test in the past 90 days

       Specific for Healthy Volunteers
   15. Physician diagnosis of asthma.

       Specific for Asthmatic Volunteers
   16. Physician directed emergency treatment for an asthma exacerbation within the preceding 3 months
   17. Moderate or Severe asthma
   18. Exacerbation of asthma more than 2x/week which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
   19. Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
   20. Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma
   21. History of intubation for asthma
   22. Use of systemic steroid therapy within the preceding 3 months for an asthma exacerbation. All use of systemic steroids in the last year will be reviewed by a study physician.
   23. Use of inhaled steroids, cromolyn or leukotriene inhibitors (Montelukast or Zafirlukast) except for use of cromolyn exclusively prior to exercise.
   24. Use of daily theophylline within the past month

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-05; Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in % neutrophils in induced sputum, comparing the 4 hr post wood smoke exposure to the baseline | baseline, and 4 hours post exposure
  Induced sputum will be collected and % neutrophils will be measured after each exposure and will be compared to baseline and each other.
Change from baseline in post wood smoke airway neutrophil influx between GSTM1 null genotype compared to GSTM1 sufficient subjects | baseline, and 4 hours post exposure
  Quantitative RT PCR will be used to measure the presence or absence of the GSTM1 transcript from blood obtained by venipuncture

SECONDARY OUTCOMES:
Change in % neutrophils in induced sputum, comparing the 24 hr post wood smoke exposure to the baseline and the change in % neutrophils from 24 hr to 4 hr post wood smoke exposure | baseline, 4 hours and 24 hours post exposure
  Induced sputum will be collected and % neutrophils will be measured after each exposure and will be compared to baseline and each other.

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, M.D., M.S., Principal Investigator — Professor
Locations (1):
- UNC Center For Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No